CLINICAL TRIAL: NCT07047599
Title: Assessment of Clinical and Uroflowmetry Parameters as Predictors of Surgical Preference in Male Patients With Lower Urinary Tract Symptoms: A Prospective Observational Study
Brief Title: Uroflowmetry and IPSS Factors Influencing Surgical Decision
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tarik Emre Sener, Assoc. Prof., Marmara University
Other Study IDs: MAR.UAD.0025
Record Dates: First submitted 2025-06-12; First posted 2025-07-02 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Lower Urinary Tract Symptom; Benign Prostate Obstruction (BPO); Voiding Dysfunction
Keywords: Lower Urinary Tract Symptoms; Benign Prostate Obstruction (BPO); Voiding Dysfunction; IPSS; Urolfowmetry
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery-Willing Group: This group includes male patients with lower urinary tract symptoms (LUTS) who indicate that they would prefer or consider surgical treatment if their symptoms remain unchanged. Participants in this group will complete the IPSS questionnaire, undergo uroflowmetry testing, and provide clinical and demographic data. No therapeutic intervention will be administered during the study.
- Non-Surgery-Willing Group: This group includes male patients with lower urinary tract symptoms (LUTS) who indicate that they do not prefer surgical treatment and would rather be followed conservatively, even if their symptoms persist. These participants will also complete the IPSS questionnaire, undergo uroflowmetry testing, and provide relevant clinical and demographic information. No therapeutic intervention will be performed.

SUMMARY:
This study aims to identify which symptoms or test findings lead men with lower urinary tract symptoms (LUTS) to consider surgical treatment. Male patients who visit the outpatient clinic for LUTS will be asked whether they would consider surgery in the future if their symptoms persist. Along with this, symptom severity scores (IPSS), quality of life scores, and uroflowmetry measurements such as maximum flow rate (Qmax) and post-void residual volume (PVR) will be collected. The goal is to determine which factors are most strongly associated with a desire for surgery. This is an observational, non-interventional study.

DETAILED DESCRIPTION:
This prospective observational study is designed to evaluate which clinical and uroflowmetry parameters are associated with a desire for surgical treatment in male patients presenting with lower urinary tract symptoms (LUTS). Participants will complete the International Prostate Symptom Score (IPSS) questionnaire, including the quality of life (QoL) item, and undergo uroflowmetry testing. Parameters such as maximum urinary flow rate (Qmax), post-void residual urine volume (PVR), and IPSS subdomain scores (e.g., weak stream, nocturia, urgency) will be analyzed. Patients will also be asked a standardized question regarding their surgical preference if their symptoms remain unchanged.

The primary aim is to determine which symptoms or objective findings (e.g., specific IPSS items, reduced Qmax) are most predictive of a preference for surgical intervention. The study will help guide clinical decision-making by identifying symptom patterns or test results that are more likely to prompt patients to consider surgery. No therapeutic intervention will be performed as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 40 years and older
* Presenting with lower urinary tract symptoms (LUTS)
* Able to complete the IPSS questionnaire
* Undergoing uroflowmetry as part of routine evaluation
* Able and willing to provide informed consent

Exclusion Criteria:

* History of urological surgery (e.g., TURP, HoLEP, radical prostatectomy)
* Presence of known prostate or bladder cancer
* Active urinary tract infection at the time of evaluation
* Neurological conditions affecting voiding (e.g., Parkinson's disease, spinal cord injury)
* Inability to perform uroflowmetry or incomplete IPSS data

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult male patients aged 40 years and older who present to the urology outpatient clinic with lower urinary tract symptoms (LUTS). All participants will complete the IPSS questionnaire and undergo uroflowmetry testing. Patients will be asked about their willingness to consider surgical treatment if their symptoms persist. No treatment or intervention will be administered as part of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Total International Prostate Symptom Score (IPSS) at Baseline | Baseline (at the outpatient clinic visit)
  Total IPSS score will be recorded for each participant at the time of initial outpatient clinic evaluation to assess symptom severity.
  Unit of Measure: Points (0 to 35)
Post-Void Residual Urine Volume (PVR) | Baseline (at the outpatient clinic visit)
  PVR will be assessed using bladder ultrasound following uroflowmetry at the initial visit.
  Unit of Measure: Milliliters (mL)
Maximum Urinary Flow Rate (Qmax) Measured by Uroflowmetry | Baseline (at the outpatient clinic visit)
  Qmax (in mL/sec) will be measured during the initial outpatient visit using non-invasive uroflowmetry.
  Unit of Measure: Milliliters per second (mL/sec)
Patient Preference for Surgery Based on a Standardized Question | Baseline (at the outpatient clinic visit)
  Patients will be asked: "Would you consider surgical treatment if your symptoms remain unchanged in the future?" Response options are Yes/No

IPD SHARING:
Plan to Share IPD: No
This study does not plan to publicly share individual participant data (IPD). However, de-identified data may be shared upon reasonable scientific request for academic or research purposes. Such requests will be evaluated on a case-by-case basis and may require institutional ethics approval and a data use agreement.